CLINICAL TRIAL: NCT01893463
Title: Prospective Study to Evaluate the Safety and Effectiveness of the iTClamp50 to Provide Temporary Wound Closure
Brief Title: Prospective Evaluation of the iTClamp50 to Provide Temporary Wound Closure
Status: Withdrawn | Type: Observational
Sponsor: Innovative Trauma Care Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-004
Record Dates: First submitted 2013-06-27; First posted 2013-07-09 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Hemorrhage; Wound Closure; Bleeding
Keywords: hemorrhage control; wound closure
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients which received the iTClamp as treatment: Use of the iTClamp50 will be determined by the EMS and ER physicians. Patients who have received treatment will be tracked from pre-hospital to patient discharge (chart review). EMS care providers and physicians will answer a survey about their experience with the iTClamp50.
  Interventions: Device: iTClamp50

INTERVENTIONS:
Device: iTClamp50

SUMMARY:
Early and effective control of severe bleeding is critical to survival of trauma patients. The iTClamp™50 is a Health Canada approved medical device for temporary wound/skin closure that quickly controls bleeding by sealing the skin. Similar to a clip, the device seals the skin edges within a pressure bar, enabling the creation of a hematoma where blood collects under pressure to form a stable clot until definitive repair. The iTClamp50 is indicated for use as a skin closure device for short-term soft tissue approximation, including use in trauma wounds, lacerations, junctional bleeds or surgical incisions. The purpose of this prospective clinical study is to evaluate the effectiveness and safety of the iTClamp50 in the ambulance (pre-hospital) and emergency department setting. This will be accomplished by observing patients with the device applied from the pre-hospital through to patient discharge. The hypothesis is that the iTClamp50 will be safe and effective at providing temporary wound closure to control hemorrhage in the pre-hospital and emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

* The device is indicated for use to control external hemorrhage from all compressible areas and to close wounds on the torso (chest and abdomen). The final decision to apply the device will be left with the care provider; however, their rationale will be reviewed in the post-use questionnaire.

Exclusion Criteria:

* The device is contraindicated for application to specific regions (e.g., eyes and genitals), application on patients less than the size of maturity, and wounds in which the skin edges cannot be approximated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pre-hospital or emergency department patients requiring wound closure for hemorrhage control
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the iTClamp50 to control hemorrhage | Patient discharge (Varies)
  As measured by length of time to control bleeding and evidence of re-bleeding
Number of Adverse Events | Until patient discharge

SECONDARY OUTCOMES:
Pain associated with application and removal of the iTClamp50 | Patient discharge (varies)
  Pain will be observed and recorded on a scale of 1-10

OTHER OUTCOMES:
Location of Application of the iTClamp50 | Immediate
  Determining where the iTClamp50 was applied (scene, ambulance, emergency department).
How long did it take for the iTClamp50 to be applied? | immediate
Anatomical Location of application of the iTClamp50 | immediate

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada